CLINICAL TRIAL: NCT06764381
Title: Study of Viral Respiratory Infections: Retrospective Evaluation of the Circulation of Respiratory Viruses, of Pathogenic-related Clinical Manifestations and of the Clinical Utility of Virological Diagnosis
Brief Title: Study of Viral Respiratory Infections
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: RESP-VIR
Record Dates: First submitted 2025-01-02; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2024-11

CONDITIONS: Respiratory Infections
Keywords: infection; virus; respiratory; RSV; SARS-CoV-2; FLUA; FLUB; AdV; MPV; PIV; Adenovirus; Metapneumovirus; Severe acute respiratory syndrome
MeSH Terms: conditions — Respiratory Tract Infections; Infections; Virus Diseases; Adenoviridae Infections; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult patients: Adult patients with request for the detection of major respiratory viruses (FLUA, FLUB, VRS, AdV, PIV, MPV, RV and SARS-CoV-2).
- Pediatric patients: Pediatric patients with request for the screening of major respiratory viruses (FLUA, FLUB, VRS, AdV, PIV, MPV, RV and SARS-CoV-2).

SUMMARY:
Acute viral respiratory infections are a major public health problem, as they cause mortality especially in pediatric patients, over 65 and those with co-morbidities. The most frequently responsible viruses are: Influenza A and B, Respiratory Syncytial Virus, Adenovirus, Parainfluenza Virus, Metapneumovirus, Rhinovirus and SARS-CoV-2. By comparing clinical data and laboratory diagnosis among all categories of patients at greatest risk, it is possible to define the symptoms associated with the pathogen and establish which etiological agents could be able to cause clinical pictures characteristics of a given type of patient. The study will also provide information on the potential role that simultaneously detected pathogens may play in determining the severity of the clinical picture. In addition, the results will allow to deepen the changes in seasonality and spread of different respiratory viruses associated with the COVID-19 pandemic.

DETAILED DESCRIPTION:
The aim of the study is:

1. Calculate the percentage of positive cases during 2018-2023.
2. Association between the viral pathogens detected individually or in packaging in respiratory material and: typology of symptomatology/clinical outcome; typology of clinical signs detectable with objective/instrumental examinations; degree of severity of clinical manifestation.
3. Reduction in the prescription of instrumental investigations (RX/ecoaddome) and reduction in the prescription of empirical antibiotic therapy with amoxicillin or amoxicillin and clavulanic acid in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult and pediatric patients, of any age, with clinical diagnosis of acute respiratory infections and with request for search of the main respiratory viruses (FLUA, FLUB, VRS, AdV, PIV, MPV, RV and SARS-CoV-2)
* Obtaining informed consent where possible.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric patients of the Sant'Orsola Hospital
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2025-02-03 (Estimated); Primary Completion 2025-03-03 (Estimated); Study Completion 2026-02-03 (Estimated)

PRIMARY OUTCOMES:
Identify potential changes in the circulation of major respiratory viruses (FLUA, FLUB, VRS, AdV, PIV, MPV, RV) during the period 2018-2023. | From 2018 to 2023
  Requests for the detection of respiratory viruses (FLUA, FLUB, VRS, AdV, PIV, MPV, RV and SARS-CoV-2) will be selected for virological diagnosis received from 2018.09.01 to 2023.08.31 and related to adult and pediatric patients at Hospitals and sampling points in the Metropolitan area of Bologna.The percentage of positive cases (positive number/ total requested) will be calculated for weeks during the study period. The comparison of the positivity found in different epidemic seasons will be performed: first (epidemic season 2018-2019), during (epidemic seasons 2019-2020, 2020-2021, 2021-2022) and after the COVID-19 pandemic (epidemic season 2022-2023) for each pathogen studied. We expect to observe differences in the frequency of each pathogen in the different weeks of the epidemic seasons 2018-2023.

SECONDARY OUTCOMES:
Define the potential role that each pathogen may have in the onset and outcome of certain clinical conditions (symptoms and clinical signs) in adult and pediatric patients | From 2022 to 2023
  The applications for virological diagnosis (FLUA, FLUB, VRS, AdV, PIV, MPV, RV and SARS-CoV-2) received during the last epidemic season (2022-2023) will be selected and relate to adult and pediatric patients of the Policlinico di S. Orsola. For each of the selected cases, data on the patient's clinical characteristics and laboratory tests will be retrieved. These data will be related to the positive findings for the viruses listed above, by means of virological diagnosis on respiratory material. In addition, the results obtained in the different categories of patients (pediatric, adult, fragile for comorbidities) will be used for the association between viral pathogens detected individually or in packaging in respiratory material and: type of symptoms/clinical outcome; type of clinical signs detectable with objective/instrumental examinations; degree of severity of the clinical manifestation.

OTHER OUTCOMES:
Assess the clinical utility of performing a correct and timely virological diagnosis in terms of reducing antibiotic therapy prescription and instrumental investigations in pediatric patients | From 2022 to 2023
  The applications for virological diagnosis (FLUA, FLUB, VRS, AdV, PIV, MPV, RV and SARS-CoV-2) received in the last epidemic season (2022-2023) and related to pediatric patients at the Policlinico di S. Orsola will be selected. For each of the selected cases, clinical and laboratory data will be retrieved. In particular, based on the diagnostic care process provided at the departments involved in the study, for patients with clinical signs that suggested the prescription of antibiotic therapy, this therapy was still prescribed, Administered only if the virus tested for is negative. For patients with factors that exposed them to risk of severe respiratory disease (age <2 years, co-morbidity) and with clinical signs that suggested the prescription of antibiotic therapy, this therapy was given and then discontinued only if the virus tested for was not found. The aim is to reduce, in pediatric patients, the prescription of instrumental investigations (RX/ecoaddome) and reduction in the pr

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Virgili, MD, Study Chair — Azienda Usl di Bologna; Maddalena Giannella, MD, Study Chair — IRCCS Azienda Ospedaliero-Universitaria di Bologna; Ilaria Corsini, MD, Study Chair — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galli C, Pellegrinelli L, Giardina F, Ferrari G, Uceda Renteria SC, Novazzi F, Masi E, Pagani E, Piccirilli G, Mauro MV, Binda S, Corvaro B, Tiberio C, Lalle E, Maggi F, Russo C, Ranno S, Vian E, Pariani E, Baldanti F, Piralla A; AMCLI-GLIViRe working group. On the lookout for influenza viruses in Italy during the 2021-2022 season: Along came A(H3N2) viruses with a new phylogenetic makeup of their hemagglutinin. Virus Res. 2023 Jan 15;324:199033. doi: 10.1016/j.virusres.2022.199033. Epub 2022 Dec 26. PMID 36581046
- [Background] Calabro GE, Rizzo C, Domnich A, DE Waure C, Rumi F, Bonanni P, Boccalini S, Bechini A, Panatto D, Amicizia D, Amodio E, Costantino C, Bert F, Lo Moro G, DI Pietro ML, Giuffrida S, Giordano V, Conversano M, Russo C, Spadea A, Ansaldi F, Grammatico F, Ricciardi R, Torrisi M, Porretta AD, Arzilli G, Scarpaleggia M, Bertola C, Vece M, Lupi C, Lorenzini E, Massaro E, Tocco M, Trapani G, Zarcone E, Munno L, Zace D, Petrella L, Vitale F, Ricciardi W. Health Technology Assessment del vaccino ricombinante adiuvato contro il virus respiratorio sinciziale (Arexvy(R)). J Prev Med Hyg. 2024 Jun 30;65(2 Suppl 1):E1-E159. doi: 10.15167/2421-4248/jpmh2024.65.2s1. eCollection 2024 Sep. No abstract available. Italian. PMID 39554593
- [Background] Piccirilli G, Rocca A, Borgatti EC, Gabrielli L, Zama D, Pierantoni L, Leone M, Totaro C, Pavoni M, Lazzarotto T, Lanari M. Respiratory Syncytial Virus-Load Kinetics and Clinical Course of Acute Bronchiolitis in Hospitalized Infants: Interim Results and Review of the Literature. Pathogens. 2023 Apr 27;12(5):645. doi: 10.3390/pathogens12050645. PMID 37242316
- [Background] De Francesco MA, Pollara C, Gargiulo F, Giacomelli M, Caruso A. Circulation of Respiratory Viruses in Hospitalized Adults before and during the COVID-19 Pandemic in Brescia, Italy: A Retrospective Study. Int J Environ Res Public Health. 2021 Sep 9;18(18):9525. doi: 10.3390/ijerph18189525. PMID 34574450